CLINICAL TRIAL: NCT01086826
Title: Neoadjuvant Docetaxel+Cisplatin and 5-fluorouracil (TPF) Followed by Radiotherapy+Concomitant Chemo or Cetuximab Versus Radiotherapy+Concomitant Chemo or Cetuximab in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck. A Randomized Phase III Factorial Study.
Brief Title: Treatment of Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Acronym: H&N07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Volontari Pazienti Oncologici (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H&N07
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RT+CDDP/5-FU (Active Comparator): RT:
  Tumor: 70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) Lymph nodes: at least 50 Gy (2 Gy x1/day, 5 days per week for 6 weeks)
  CDDP: 20 mg/m2/day as 30 minutes IV infusion from day 1 to day 4 5-FU 800 mg/m2/day for 4 will be administered as continuos iv infusion Both drugs will be administered during weeks 1 and 6 of irradiation, starting from day 1 of radiotherapy.
  Interventions: Drug: RT+CDDP/5-FU
- RT+CETUXIMAB (Experimental): RT:
  Tumor: 70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) Lymph nodes: at least 50 Gy (2 Gy x1/day, 5 days per week for 6 weeks)
  CETUXIMAB:
  Cetuximab 400 mg/m2 as first dose, 7 days before the beginning of radiotherapy as 120 minutes IV infusion. Subsequent doses of 250 mg/ m2 will be administered as 60 minutes IV infusion, weekly, for 7 times.
  Interventions: Drug: RT+CETUXIMAB
- INDUCTION CTx(TPF)+(RT+CDDP/5-FU) (Active Comparator): INDUCTION CTx(TPF):
  DOCETAXEL:
  75 mg/m², 1 hour IV infusion, Day and every 3 weeks
  CISPLATIN:
  80mg/m², intravenous infusion over 30-minute to 3 hours,Day 1 immediately after docetaxel administration and then every 3 weeks 5-FU 800 mg/m²/day, 24 hour continous infusion over 4 days, Day 1 after the end of cisplatin infusion, and every 3 weeks.
  RT:
  Tumor: 70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) Lymph nodes: at least 50 Gy (2 Gy x1/day, 5 days per week for 6 weeks)
  CDDP: 20 mg/m2/day as 30 minutes IV infusion from day 1 to day 4 5-FU 800 mg/m2/day for 4 will be administered as continuos iv infusion
  Interventions: Drug: INDUCTION CTx(TPF)+(RT+CDDP/5-FU)
- INDUCTION CTx(TPF)+(RT+CETUXIMAB) (Experimental): DOCETAXEL:
  75 mg/m², 1 hour IV infusion, Day and every 3 weeks
  CISPLATIN:
  80mg/m², intravenous infusion over 30-minute to 3 hours,Day 1 immediately after docetaxel administration and then every 3 weeks 5-FU 800 mg/m²/day, 24 hour continous infusion over 4 days, Day 1 after the end of cisplatin infusion, and every 3 weeks.
  RADIOTHRAPY:
  Tumor: 70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) Lymph nodes: at least 50 Gy (2 Gy x1/day, 5 days per week for 6 weeks)
  CETUXIMAB:
  Cetuximab 400 mg/m2 as first dose, 7 days before the beginning of radiotherapy as 120 minutes IV infusion. Subsequent doses of 250 mg/ m2 will be administered as 60 minutes IV infusion, weekly, for 7 times.
  Interventions: Drug: INDUCTION CTx(TPF)+(RT+CETUXIMAB)

INTERVENTIONS:
Drug: RT+CDDP/5-FU — RT=70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) CDDP: 20 mg/m2/day as 30 minutes IV infusion from day 1 to day 4 5-FU: 800 mg/m2/day for 4 days Both drugs will be administered during weeks 1 and 6 of irradiation, starting from day 1 of radiotherapy.
  Other Names: Radiotherapy, Cisplatin, 5-fluoruracil
  Arms: RT+CDDP/5-FU
Drug: RT+CETUXIMAB — RT= 70 Gy (2 Gy x1/day, 5 days per week for 7 weeks) Cetuximab= 400 mg/m2 as first dose.Subsequent doses of 250 mg/ m2, weekly, for 7 times.
  Other Names: Radiotherapy, Cetuximab
  Arms: RT+CETUXIMAB
Drug: INDUCTION CTx(TPF)+(RT+CDDP/5-FU) — INDUCTION CTx(TPF):docetaxel 75 mg/m² + CDDP 80mg/m² + 5-FU 800 mg/m²/day from day 1 to day 4 will begin after the end of cisplatin infusion on day 1.Every 3 weeks.
  concomitant CTx= CDDP 20 mg/m2/day + 5-FU 800 mg/m2/day RT= 70 Gy(2 Gy x1/day, 5 days per week for 7 weeks)
  Other Names: Docetaxel. Cisplatin, 5-fluoruracil, Radiotherapy
  Arms: INDUCTION CTx(TPF)+(RT+CDDP/5-FU)
Drug: INDUCTION CTx(TPF)+(RT+CETUXIMAB) — INDUCTION CTx(TPF):docetaxel 75 mg/m² + CDDP 80mg/m² + 5-FU 800 mg/m²/day from day 1 to day 4 will begin after the end of cisplatin infusion on day 1.Every 3 weeks.
  RT= 70 Gy(2 Gy x1/day, 5 days per week for 7 weeks) CETUXIMAB= 400 mg/m2 as first dose. Subsequent doses of 250 mg/ m2, weekly, for 7 times.
  Other Names: Docetaxel. Cisplatin, 5-fluoruracil, Radiotherapy, Cetuximab
  Arms: INDUCTION CTx(TPF)+(RT+CETUXIMAB)

SUMMARY:
This is a randomized multicenter open label phase III factorial trial evaluating the 3 years OS in patients with locally advanced squamous cell carcinoma of head and neck treated with locoregional treatment (radiotherapy plus concomitant chemotherapy or cetuximab) with or without neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This multicenter open label randomised phase III study is the implementation of a previous phase II randomized trial evaluating the efficacy of chemoradiotherapy with or without neoadjuvant TPF chemotherapy in locally advanced Head and Neck cancer. Assuming a randomisation ratio of 1:1, using the Mantel-Cox version of the log-rank test, 204 events are required in order to achieve a power of 0.80 of detecting an hazard ratio of 0.675 in favour of the experimental treatment with a type I error of 0.05, two-sided. With a uniform accrual of 4 years and a follow-up of 2 further years, the total number of required patients is 420 (210 per arm) to detect an absolute difference of 12% in 3 year overall survival in favour of the neoadjuvant arm (from 52.5% to 64.5%).Since the 101 patients randomized in the phase II part of the study will be included in the final analysis, 319 new patients are needed to complete the trial.The total number of 420 patients will be able to detect a difference of 10%, (from 35% to 45%) in terms of grade 3/4 in-field mucosal toxicity during the concomitant treatment (radiotherapy plus chemo or cetuximab) with a power of 80%. Within the H&N07 trials was introduced a sub-study that allows to investigate the value of circulating marker evaluation as predictor of response to anti EGFR therapy in patients with cancer of the head and neck.

The expression level analysis of circulating biological markers will be evaluated on blood collected during therapy. The analysis will concern the following biological markers:Cytokines angiogenesis and cell adhesion molecules; Proteins involved in the EGFR signaling pathway (EGF, TGF-a, s-EGFR);circulating tumor cells (CTC) and circulating endothelial cells (CEC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven squamous cell carcinoma of the head and neck.
2. Primary tumor sites eligible : oral cavity, oropharynx, hypopharynx Although they are admittedly of squamous cell types, the following tumors will be excluded because of them responsiveness to chemotherapy: tumors of the nasal and paranasal cavities and of the nasopharynx.
3. Stage 3 or 4 disease without evidence of distant metastases verified by chest X Ray, abdominal ultrasound, or CT (liver function test abnormalities); bone scan in case of local symptoms.
4. At least one uni or bidimensionally measurable lesion.
5. Tumor considered inoperable after evaluation by a multidisciplinary team (i.e. a surgeon, a medical oncologist and a radiation oncologist). Criteria for inoperability are:

   1. technical unresectability: tumor fixation/invasion to base of the skull or cervical vertebrae, involvement of the nasopharynx, and fixed lymph nodes.
   2. Physician decision based on low surgical curability. This category will include the following:

   i) All T3-4 stages. ii) All N2-3 stages excluding T1 N2. iii) Patients for organ preservation. Reason for inoperability will be recorded in the CRF.
6. No previous chemotherapy or radiotherapy for any reason and no previous surgery for SCCHN (other than biopsy) are allowed at time of study entry.
7. Age > 18 years.
8. Karnofsky performance status > 70. (ECOG 0-1) (Appendix II)
9. No active alcohol addiction.
10. Life expectancy > 6 months.
11. Signed informed consent prior to beginning protocol specific procedures.
12. Adequate bone marrow, hepatic and renal functions as evidenced by the following:

    a) Hematology (Bone marrow): i) Neutrophils > 2.0 109/L ii) Platelets > 100 x 109/L iii) Hemoglobin > 10 g/dL b) Hepatic function i) Total bilirubin < 1 x UNL ii) ASAT (SGOT) and ALAT (SGPT) < 2.5 x ULN iii) Alkaline phosphatase < 5 x ULN Patients with ASAT or ALAT > 1.5 x ULN associated with alkaline phosphatase > 2.5 x ULN are not eligible for the study.

    c) Renal function : serum creatinine < 1 x UNL. In case of borderline value the creatinine clearance > 60 ml/min (calculated by the Cockcroft-Gault method as follows :
13. Patients must be available for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating center.

    -

Exclusion Criteria:

1. Pregnant or lactating women or women of childbearing potential not using adequate contraception.
2. Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin, or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years. Any prior treatment with radiotherapy or chemotherapy is an exclusion criterion.
3. Symptomatic peripheral neuropathy > grade 2 by NCIC-CTG criteria
4. Symptomatic altered hearing > grade 2 by NCIC-CTG criteria.
5. Other serious illnesses or medical conditions including:

   1. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry.
   2. History of significant neurologic or psychiatric disorders including dementia or seizures.
   3. Active uncontrolled infection.
   4. Active peptic ulcer.
   5. Hypercalcemia.
   6. Chronic obstructive pulmonary disease requiring hospitalization during the year preceding study entry
6. History of hypersensitivity reaction to polysorbate 80 (Appendix IV)
7. Patients requiring intravenous alimentation.
8. Patients who experienced a weight loss of more than 20% of their body weight in the 3 months preceding study entry.
9. Concomitant treatment with any other anticancer therapy.
10. Participation in a therapeutic clinical trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-03; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years
  overall survival defined as the time from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
progression free survival | 3 years
  Secondary Objectives are: To compare the radiological and pathological complete response rate, the duration of response,the time to progression,the hematological and non-hematological toxicity,the duration of RTX plus concomitant CHT or cetuximab,the interruption number and the radiological complete response during concomitant chemoradiation and radiation plus cetuximab. To evaluate the biological profile expression,correlation between biological biomarkers expression,response to treatment and OS. To compare Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Ghi, MD, Principal Investigator — Ospedale SS Giovanni e Paolo - Venezia, Italy
Locations (60):
- Italy (60):
  - Istituto tumori "Giovanni Paolo II" IRCCS, Bari, Bari
  - Ospedale S.Martino, Belluno, Belluno
  - Ospedale "S. Maria Del Prato", Feltre, Belluno
  - Ospedale Di Treviglio - Caravaggio, Treviglio, Bergamo
  - Ospedale Bellaria Di Bologna, Bologna, Bologna
  - Policlinico S.Orsola-Malpighi, Bologna, Bologna
  - Ospedale "S.Maurizio", Bolzano, Bolzano
  - Istituto Clinico S.Anna, Brescia, Brescia
  - "Ospedale Businco", Cagliari, Cagliari
  - Policlinico Universitario, Cagliari, Cagliari
  - A.O Pugliese-Ciaccio, Catanzaro, Catanzaro
  - Ospedale Clinicizzato Di Chieti, Chieti, Chieti
  - A.O. Ospedale Sant'Anna, S.Fermo, Como
  - Ospedale "AUGUSTO MURRI", Fermo, Fermo
  - A.O.Universitaria, Ferrara, Ferrara
  - IRCCS Casa Sollievo della Sofferenza, S. Giovanni Rotondo, Foggia
  - Azienda Ospedaliera "Alessandro Manzoni", Lecco, Lecco
  - Ospedale di Macerata, Macerata, Macerata
  - Ospedale "B.Eustachio" - S.Severino, San Severino Marche, Macerata
  - P.O. SAN VINCENZO di Messina, Messina, Messina
  - A.O. Universitaria Di Messina, Messina, Messina
  - Irccs - Ospedale "S. Raffaele", Milan, Milano
  - "Istituto Europeo di Oncologia", Milan, Milano
  - "Ospedale San Paolo", Milan, Milano
  - A.O. Niguarda-Cà Granda, Milan, Milano
  - "A.O. - Policlinico Di Modena", Modena, Modena
  - H.S. Gerardo dei Tintori, Monza, Moza-Brianza
  - Ospedale Di Camposampiero, Camposampiero, Padova
  - Ospedale Civile di Cittadella, Cittadella, Padova
  - "Istituto Oncologico Veneto", Padua, Padova
  - Policlinico Universitario di Palermo, Palermo, Palermo
  - Casa di Cura "La Maddalena", Palermo, Palermo
  - A.O.Universitaria "Ospedale Maggiore", Parma, Parma
  - Osp. S. Maria della Misericordia, Perugia, Perugia
  - Ospedale Santa Croce Di Fano, Fano, Pesaro-urbino
  - A.O. "Ospedale S. Salvatore", Pesaro, Pesaro-urbino
  - Ospedale "G. Da Saliceto", Piacenza, Piacenza
  - Osp. S. Maria Delle Croci, Ravenna, Ravenna
  - A.O. "S.Camillo de' Lellis", Rieti, Rieti
  - Istituto Nazionale Tumori Regina Elena, Roma, Roma
  - Ospedale S.Pietro "Fatebenefratelli", Roma, Roma
  - Ospedale Civile Di Sondrio, Sondrio, Sondrio
  - Osp. S.G. Moscati, Taranto, Taranto
  - Ospedale "S. Chiara", Trento, Trento
  - Ospedale Civile di Castelfranco, Castelfranco Veneto, Treviso
  - Ospedale Ca' Foncello, Treviso, Treviso
  - "Ospedali Riuniti", Trieste, Trieste
  - Ospedale Civile di Latisana, Latisana, Udine
  - P.O. "S.Antonio Abate", Tolmezzo, Udine
  - A.O. Santa Maria della Misericordia, Udine, Udine
  - Azienda Ospedaliera Di Circolo, Busto Arsizio, Varese
  - Azienda Ospedaliera "S.Antonio Abate", Gallarate, Varese
  - Ospedale Di Circolo E Fondazione Macchi, Varese, Varese
  - "Ospedale dell' Angelo", Mestre, Venezia
  - "Ospedale Civile di Mirano", Mirano, Venezia
  - Ospedale Civile SS Giovanni e Paolo, Venezia, Venezia
  - "AULSS 21 Mater Salutis", Legnago, Verona
  - Ospedale Civile Maggiore Borgo Trento, Verona, Verona
  - Ospedale "Boldrini", Thiene, Vicenza
  - Ospedale civile di Vicenza, Vicenza, Vicenza

REFERENCES:
- [Derived] Ghi MG, Paccagnella A, Ferrari D, Foa P, Alterio D, Codeca C, Nole F, Verri E, Orecchia R, Morelli F, Parisi S, Mastromauro C, Mione CA, Rossetto C, Polsinelli M, Koussis H, Loreggian L, Bonetti A, Campostrini F, Azzarello G, D'Ambrosio C, Bertoni F, Casanova C, Emiliani E, Guaraldi M, Bunkheila F, Bidoli P, Niespolo RM, Gava A, Massa E, Frattegiani A, Valduga F, Pieri G, Cipani T, Da Corte D, Chiappa F, Rulli E; GSTTC (Gruppo di Studio Tumori della Testa e del Collo) Italian Study Group. Induction TPF followed by concomitant treatment versus concomitant treatment alone in locally advanced head and neck cancer. A phase II-III trial. Ann Oncol. 2017 Sep 1;28(9):2206-2212. doi: 10.1093/annonc/mdx299. PMID 28911070